CLINICAL TRIAL: NCT02795871
Title: Multicentric Evaluation of in Utero Dexamethasone (DEX) on the Cognitive Development of Children at Risk of Congenital Adrenal Hyperplasia
Brief Title: Prenatal Dex Study
Acronym: Prenatal Dex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL14_0447
Record Dates: First submitted 2016-05-25; First posted 2016-06-10 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; Prenatal treatment; Dexamethasone; Neuropsychological assessment; Cognitive development
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group D+ 1 (Experimental): Girls and boys at risk of CAH treated in utero by Dexamethasone but unaffected.
  Interventions: Behavioral: Neuropsychological and cognitive assessment
- Group D+ 2 (Experimental): Girls and boys affected by CAH and treated in utero by Dexamethasone.
  Interventions: Behavioral: Neuropsychological and cognitive assessment
- : Group D - 1 (Active Comparator): Girls and boys not affected by CAH and not treated in utero by Dexamethasone.
  Interventions: Behavioral: Neuropsychological and cognitive assessment
- Group D - 2 (Active Comparator): Girls and boys affected by CAH and not treated in utero by Dexamethasone.
  Interventions: Behavioral: Neuropsychological and cognitive assessment
- Group D - 3 (Other): Girls and boys enrolled in school closed to Lyon
  Interventions: Behavioral: Neuropsychological and cognitive assessment

INTERVENTIONS:
Behavioral: Neuropsychological and cognitive assessment

SUMMARY:
The classic form of 21-hydroxylase deficiency (prevalence 1/15,000) is the most common cause of congenital adrenal hyperplasia (CAH). This autosomic recessive disease is responsible for virilization of the external genitalia in girls through androgen hypersecretion during fetal life. Since 1984, the Lyon Pediatric Endocrinology group has proposed prenatal dexamethasone (DEX) for all fetuses at risk of CAH With the aim of preventing fetal androgen hypersecretion in affected girls and avoiding poor long-term results from reconstructive surgery. Prenatal DEX was used in Europe and the USA but its use was recently suspended: in 2007, a Swedish study conducted on 26 children treated with DEX in utero for a short period of time reported cognitive impairments. These data were not confirmed by an American study on the short-term DEX use, which showed potential cognitive impairments in CAH children exposed to DEX for long periods of time. These confusing and controversial results have caused the scientific community to question its position and have resulted in the suspension of the use of prenatal DEX with drastic consequences for CAH girls (virilization; genital surgery etc.). In this context, an evaluation of neuropsychological development under in utero DEX is essential to validate its indication for use during the prenatal period. This study will evaluate outcomes using prospective cognitive and emotional assessments. It will first focus on the unaffected children previously treated in utero in order to assess the adverse effects of the drug. The study will then assess the children with CAH for whom DEX could have beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

Groups D+1, D+2, D-1 and D-2

* Male or female
* Patient with Congenital Adrenal Hyperplasia or sibling of a CAH patient
* Age: 6 to 15 years (at the time of inclusion)
* The subject's legal representatives have understood the information note/informed consent form, obtained answers to all their questions and have given signed, written, informed consent
* Subject with health insurance

Group D-3 (Schoolchildren)

* Male or female
* With no connection with Congenital Adrenal Hyperplasia
* Age: 6 to 15 years (at the time of inclusion)
* The subject's legal representatives have understood the information note/informed consent form, obtained answers to all their questions and have given signed, written, informed consent
* Subject with health insurance

Exclusion Criteria:

For all groups :

* Patient/Subject with another genetic disease
* Patient/Subject with known neuropsychology disease(s)
* Patient/Subject whose mother has received another treatment during her pregnancy with possible known adverse events on the neuropsychological development of the child

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Intelligence quotient | 3 months
  Wechsler Intelligence Scale for Children (WISC) is designed to measure human intelligence. WISC-IV includes:
  * Verbal Comprehension Index: measure of verbal concept formation.
  * Perceptual Reasoning Index: measure of non-verbal and fluid reasoning.
  * Working Memory Index: measure of working memory.
  * Processing Speed Index: measure of processing speed. Data measured: raw score (0 to 150), standard score (1 to 19), index (40 to 160).
  The four indexes of the intelligence quotient will be considered hierarchically as follows: first the Working Memory Index, then the Processing Speed Index, third the Perceptual Reasoning Index, fourth the Verbal Comprehension Index.

SECONDARY OUTCOMES:
Children Memory Scale (CMS) | 3 months
  Neurocognitive profile of children assessed by Children Memory Scale (CMS) at Visit 2.
  Memory tests: Children Memory Scale (CMS), the following composites will be considered in our study:
  * Immediate and delayed visual memory : face recognition and dot location
  * Immediate and delayed verbal memory, recognition : stories, word pairs
  * Learning: dot location and word pairs
  * Attention, concentration: numbers, sequences
Rey figure test | 3 months
  Neurocognitive profile of children assessed by visuoperceptual test (Rey Figure test) at Visit 2
Revised - Child Measure of Anxiety Scale (R- CMAS) score | 15 months
  Emotional profile assessed by Revised - Child Measure of Anxiety Scale (R- CMAS) score
Mood Depressive Inventory for Children (MDI- C) score | 15 months
  Emotional profile assessed by Mood Depressive Inventory for Children (MDI- C) score
Child Behavior Checklist (CBCL) score | 15 months
  Emotional profile assessed by Child Behavior Checklist (CBCL) score
Evaluation of the benefits of in utero DEX in preventing or reducing the virilization of external genitalia in CAH girls | Day 1
  The anatomical evaluation (phenotyping) of girls' external genitalia was performed at the time of the surgical correction and included the measurement of the genital tubercule (GT), the distance between the perineum and the urethra-vaginal confluence, the degree of fusion of the genital folds (labia majora), their pigmentation and creases. The measurement of the ano-genital distance was not routine practice in the past.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique TARDY-GUIDOLLET, MD PHD, Principal Investigator — Groupement Hospitalier Est - Laboratoire d'endocrinologie moléculaire et maladies rares - Centre de biologie et de pathologie Est.
Locations (10):
- France (10):
  - Service d'endocrinologie pédiatrique, CHU de Besançon, Besançon
  - Service d'endocrinologie pédiatrique, CHU de Bordeaux, Bordeaux
  - Groupement Hospitalier Est - Laboratoire d'endocrinologie moléculaire et maladies rares - Centre de biologie et de pathologie Est. 59 boulevard Pinel, Bron
  - Service d'endocrinologie pédiatrique, CHU de Grenoble, Grenoble
  - Service d'endocrinologie pédiatrique, CHRU de Lille, Lille
  - Service d'endocrinologie pédiatrique, Hopital de la Timone, APHM, Marseille
  - Service d'endocrinologie pédiatrique, CHU de Nantes, Nantes
  - Service d'endocrinologie pédiatrique, CHU de Nice, Nice
  - Service d'endocrinologie pédiatrique, Hôpital Armand Trousseau, AP-HP, Paris
  - Service d'endocrinologie pédiatrique, CHU de Reims, Reims